CLINICAL TRIAL: NCT06798467
Title: An in Vivo "Evaluation of Post Obturation Pain Associated With Calcium Hydroxide-based Root Canal Sealers and Resin-based Root Canal Sealer: a Single Visit Root Canal Treatment
Brief Title: Evaluation of Post Obturation Pain Associated With Calcium Hydroxide-based Root Canal Sealers and Resin-based Root Canal Sealer: a Single Visit Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Sindh Medical University (Other)
Responsible Party: Principal Investigator, Soha Pirzado, BDS, FCPS-II TRAINEE, Jinnah Sindh Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JSMU/IRB/2024/971
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Root Canal Sealers; Post Operative Pain; Irreversible Pulpitis
Keywords: root canal sealers; post operative pain; symptomatic periapical periodontitis; calcium hydroxide sealer; resin-based root canal sealer; visual analogue scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- post obturation pain (Active Comparator): Unpleasant sensation of any degree of pain after root canal treatment.
  Interventions: Other: Endodontic sealer
- endodontic sealer (Active Comparator): endodontic sealer is a material used in root canal therapy to fill the microscopic spaces between the root canal filling material (typically gutta-percha) and the walls of the root canal. Its primary function is to create a tight seal that prevents the ingress of bacteria and fluids into the root canal system, helping to prevent reinfection and promoting the healing of periapical tissues. Endodontic sealers also help to ensure that the root canal filling reaches all parts of the canal, especially in complex or irregularly shaped anatomies.
  Interventions: Other: post obturation pain

INTERVENTIONS:
Other: Endodontic sealer — endodontic sealer is a material used in root canal therapy to fill the microscopic spaces between the root canal filling material (typically gutta-percha) and the walls of the root canal. Its primary function is to create a tight seal that prevents the ingress of bacteria and fluids into the root canal system, helping to prevent reinfection and promoting the healing of periapical tissues. Endodontic sealers also help to ensure that the root canal filling reaches all parts of the canal, especially in complex or irregularly shaped anatomies.
  Arms: post obturation pain
Other: post obturation pain — Unpleasant sensation of any degree of pain after root canal treatment.
  Arms: endodontic sealer

SUMMARY:
The objective of this study is to evaluate the post obturation pain associated with calcium hydroxide-based root canal sealer and resin-based root canal sealer after single visit root canal treatment following endodontic treatment by means of Visual Analog Scale.

Methods: This study was designed as single blind, randomized control trial. Sixty patients with irreversible pulpitis requiring endodontic canal treatment were recruited by probability random sampling into two groups based on root canal sealer used during endodontic treatment: calcium hydroxide-based root canal sealer and resin-based root canal sealer . The post-operative pain of patients was recorded via a telephone call at 6 hours, 24 hours, and at 48hours on the visual analogue scale (VAS).

DETAILED DESCRIPTION:
Modern endodontics offers advancements in technologies, procedures and materials. Post-obturation pain is defined as pain of any degree that occurs after initiation of root canal treatment1 and its occurrence was noted to vary between 3 and 58%.2 3 The causes of postoperative pain is related to post obturation pain and can be classified as mechanical, chemical and/or microbiological injuries to the peri-radicular tissues.Factors identified that contribute to post-operative pain after single- visit root canal treatment consist of the following: age, sex, tooth type or location. Intraoperative factors include the physical properties of endodontic instruments used in the initial treatment, features of irrigation protocol like chemical solutions and concentrations, microbiological stability and resistance, histopathological state of the tissues surrounding the tooth, etc.6 During the obturation phase of root canal therapy, the endodontic sealer makes direct and local contact with the reshaped periapical tissues through the apical foramen and any supplementary lateral canals. By understanding the factors that contribute to postoperative pain, dental practitioners may better choose procedures and supplies that have been shown to reduce the occurrence of this symptom.7 Pain perception is mainly a subjective and variable experience that depends on many psychological and physical factors. The visual analog scale (VAS) is usually used as a measure of pain intensity in clinical researches due to its simplicity. The VAS intensity rating consisted of a 100-mm length line with two end points as no pain and worst pain. 8 An ideal root canal sealer should be capable of creating an effective bond to the GP and root canal walls to prevent microleakage at the interface.9 Biocompatibility and bioactivity are essential properties for root canal sealers, as these materials are in close proximation with the surrounding tissues and affect the repair.10 If the sealers are biocompatible and soluble in tissue fluid, minimal extrusions could be tolerated by the peri-radicular tissues.11 Sealers placed in the root canals interfere with periodontal tissues through the apical foramina, lateral canals, or leaching and can potentially affect the healing process in the periodontium Thus, the local inflammation caused by root canal obturation materials may result in postoperative pain. The intensity of inflammatory reactions depends on a number of different factors, including the composition of the sealer. 12 Therefore, root canal sealers may have a role in the discomfort felt after having a root canal. Pain sensations and flare-ups may be triggered by root canal sealers due to the stimulation of trigeminal nociceptors in vitro and the accompanying immunologic response, as proposed by Ruparel et al13 The un-polymerized residues remain due to formation of oxygen inhibition layer in the mixture of AH Plus sealer, which is responsible for maintaining its toxic effect.14 Sealapex is one of calcium hydroxide based root canal sealer having cytotoxic potential. After setting Sealapex becomes unstable and disintegrates.15 Khatri S1 in his study stated that AH Plus was associated with the highest pain intensity post 12 hours evaluation 5.00±1.124. This signifies the increased toxic effect of AH Plus sealer then Sealapex. AH Plus contains both epoxy resins and amines which have toxic effect. A randomized controlled clinical investigation by Ates et al16 including both vital and non-vital mandibular premolars and molars found a 68% and 59% prevalence of patients experiencing discomfort in teeth filled with AH Plus sealer.

The aim of this in-vivo study is to compare and evaluate the effect of AH Plus and Sealapex sealers on postoperative pain. Given the conflicting findings and lack of data in the endodontic literature on this issue, we decided to investigate the connection between endodontic sealers and postoperative discomfort. The purpose of this randomized clinical trial was to evaluate the effectiveness of two root canal sealer AH Plus and sealapex in reducing postoperative pain and the need for analgesics following root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients presenting with signs and symptoms of irreversible pulpitis in maxillary or mandibular teeth

  * ≥18 years of age.

Exclusion Criteria:

* • Patients with any systemic diseases

  * Retreatment cases
  * Teeth with calcified canals.
  * Medically compromised patient (with immunosuppressive/ systemic diseases, patient on medication)
  * Patients on analgesics or sedative medication prior to root canal therapy.
  * Patients in whom single visit endodontic treatment will not be possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of post obturation pain associated with calcium hydroxide-based root canal sealers and resin-based root canal sealer: a single visit root canal treatment. | 6 hours, 24 hours and 48 hours
  Introduction: Modern endodontics offers advancements in technologies, procedures and materials. Post-obturation pain is defined as pain of any degree that occurs after initiation of root canal treatment and its occurrence was noted to vary between 3 and 58%. The objective is to evaluate the post obturation pain associated with calcium hydroxide-based root canal sealer and resin-based root canal sealer after single visit root canal treatment following endodontic treatment by means of Visual Analog Scale.
  Methods: This study was designed as single blind, randomized control trial .Sixty patients with irreversible pulpitis requiring endodontic canal treatment were recruited by probability random sampling into two groups based on irrigation protocols used during endodontic treatment: calcium hydroxide-based rootand resin-based root canal sealer . The post-operative pain of patients was recorded via a telephone call at 6 hours, 24 hours, and at 48 hours on the visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Sindh Institute of Oral Health Sciences Jinnah Sindh Medical University Karachi, Karcahi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Khatri S, Parvez S, Agarwal MK, Goyal D, Binawra KK, Jain A, et al. Comparative Evaluation of Effect of Resinbased, Calcium Hydroxide-Based and Bioceramic-Based Root Canal Sealers on Postoperative Pain. List of Articles Pages No.2022;11(1) :54-61